CLINICAL TRIAL: NCT00661362
Title: A 24-Week International, Multi-centre, Randomized, Parallel-group, Double-blind, Placebo-Controlled, Phase III Study to Evaluate the Efficacy and Safety of Saxagliptin in Combination With Metformin in Adult Patients With Type 2 Diabetes Who Have Inadequate Glycaemic Control on Metformin Therapy
Brief Title: Evaluate Efficacy and Safety of Saxagliptin in Combination With Metformin in Adult Patients With Type 2 Diabetes
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Collaborators: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: D1680C00006
Record Dates: First submitted 2008-04-17; First posted 2008-04-18 (Estimated); Results first posted 2012-03-08 (Estimated); Last update posted 2012-03-08 (Estimated); Status verified 2012-02

CONDITIONS: Type 2 Diabetes
Keywords: DPP-4 inhibitors; HbA1c; Incretins
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — saxagliptin; Metformin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Experimental): Metformin + Saxagliptin
  Interventions: Drug: Saxagliptin; Drug: Metformin
- 2 (Placebo Comparator): Metformin + Placebo
  Interventions: Drug: Placebo; Drug: Metformin

INTERVENTIONS:
Drug: Saxagliptin — Oral tablet, once daily for 24 weeks
  Other Names: Onglyza
  Arms: 1
Drug: Placebo — oral tablet, once daily for 24 weeks
  Arms: 2
Drug: Metformin — oral tablet, once daily for 24 weeks
  Other Names: Glucophage

SUMMARY:
Saxagliptin is a new investigational medication being developed for treatment of type 2 diabetes. This study is designed to evaluate the efficacy and safety in adult patients who have inadequate glycaemic control when treated with metformin in addition to diet and exercise.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with Type 2 diabetes
* Treatment with metformin at a stable dose >1500 mg/day
* HbA1c ≥ 7.0% and ≤10.0%

Exclusion Criteria:

* Insulin therapy within one year of enrolment (with the exception of insulin therapy during a hospitalization or use in gestational diabetes)
* Type 1 diabetes, history of ketoacidosis, or hyperosmolar non-ketonic koma

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 570 (Actual)
Dates: Start 2008-06; Primary Completion 2009-09 (Actual); Study Completion 2009-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Peter Ohman, MD, Study Director — AstraZeneca; Deborah Price, MSc, Study Chair — AstraZeneca
Locations (30):
- China (16):
  - Research Site, Hefei, Anhui
  - Research Site, Beijing, China
  - Research Site, Chongqing, China
  - Research Site, Guangzhou, Guangdong
  - Research Site, Shijiazhuang, Hebei
  - Research Site, Ha'er Bing, Hei Longjiang
  - Research Site, Wuhan, Hubei
  - Research Site, Changsha, Hunan
  - Research Site, Nanjing, Jiangsu
  - Research Site, Changchun, Jilin
  - Research Site, Dalian, Liaoning
  - Research Site, Shenyang, Liaoning
  - Research Site, Shanghai, Shanghai Municipality
  - Research Site, Chengdu, Sichuan
  - Research Site, Hangzhou, Zhejiang
  - Research Site, Tianjin
- India (5):
  - Research Site, Hyderabad, Andhra Pradesh
  - Research Site, Bangalore, Karnataka
  - Research Site, Mangalore, Karnataka
  - Research Site, Nagpur, Maharashtra
  - Research Site, Bangalore
- South Korea (9):
  - Research Site, Seongnam-si, Gyeonggi-do
  - Research Site, Bucheon-si
  - Research Site, Daegu
  - Research Site, Goyang
  - Research Site, Gwangju
  - Research Site, Incheon
  - Research Site, Pusan
  - Research Site, Seoul
  - Research Site, Uijeongbu-si

REFERENCES:
- [Derived] Perl S, Cook W, Wei C, Iqbal N, Hirshberg B. Saxagliptin Efficacy and Safety in Patients With Type 2 Diabetes and Moderate Renal Impairment. Diabetes Ther. 2016 Sep;7(3):527-35. doi: 10.1007/s13300-016-0184-9. Epub 2016 Jul 11. PMID 27402391
- [Derived] Yang W, Pan CY, Tou C, Zhao J, Gause-Nilsson I. Efficacy and safety of saxagliptin added to metformin in Asian people with type 2 diabetes mellitus: a randomized controlled trial. Diabetes Res Clin Pract. 2011 Nov;94(2):217-24. doi: 10.1016/j.diabres.2011.07.035. Epub 2011 Aug 26. PMID 21871686

RESULTS

PARTICIPANT FLOW:
Groups:
- Saxagliptin 5 mg + Metformin: Saxagliptin 5 mg tablet, once daily (OD), added on to stable Metformin for 24 weeks
- Placebo + Metformin: Placebo tablet, OD, added on to stable Metformin for 24 weeks
Period: Overall Study
Arm/Group | Saxagliptin 5 mg + Metformin | Placebo + Metformin
Started | 283 (Randomized and treated) | 287 (Randomized and treated)
Completed | 254 (Completed 24 Weeks of treatment) | 247 (Completed 24 Weeks of treatment)
Not Completed | 29 | 40
Not completed — Adverse Event | 5 | 4
Not completed — Incorrect enrollment | 2 | 0
Not completed — Study specific discontinuation criteria | 4 | 11
Not completed — Withdrawal by Subject | 13 | 23
Not completed — Lost to Follow-up | 3 | 1
Not completed — Severe non-compliance to protocol | 0 | 1
Not completed — Safety reasons | 1 | 0
Not completed — Metformin dose haven't decreasd to 2.5 g | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Saxagliptin 5 mg + Metformin | Placebo + Metformin | Total
Number analyzed (Participants) | 283 | 287 | 570
Age Continuous [Mean (Standard Deviation); unit: Years] | 53.75 (10.42) | 54.36 (10.06) | 54.05 (10.24)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 147 | 148 | 295
  Male | 136 | 139 | 275

OUTCOME MEASURES:

1. Primary Outcome: Absolute Change From Baseline to Week 24 in Glycosylated Haemoglobin A1c (HbA1c)
Description: Adjusted* mean change from baseline in HbA1c achieved with saxagliptin 5 mg + metformin versus placebo + metformin at week 24 (LOCF, Full Analysis set). HbA1c is a continuous measure, the change from baseline for each subject is calculated as the week 24 values minus the baseline value. *Adjusted for baseline HbA1c.
Time Frame: Baseline , Week 24
Population: Randomized participants who took at least 1 dose of double-blind treatment. To be included in analysis: change from baseline to Wk 24 LOCF for efficacy, subjects must have had a baseline and at least 1 post baseline efficacy measurement.
Measure: Mean (Standard Error); unit: percent
Arm/Group | Saxagliptin 5 mg + Metformin | Placebo + Metformin
Number analyzed (Participants) | 275 | 279
percent
  Baseline | 7.90 (0.049) | 7.94 (0.050)
  Week 24 | 7.10 (0.056) | 7.55 (0.062)
  adjusted baseline HbA1c | -0.78 (0.051) | -0.37 (0.050)
Statistical Analysis 1: Comparison: Saxagliptin 5 mg + Metformin vs Placebo + Metformin; Test type: Superiority or Other; p < 0.0001, ANCOVA; Mean Difference (Net) = -0.42, 95% CI 2-sided [-0.55 to -0.29], Standard Error of Mean 0.067

2. Secondary Outcome: Absolute Change From Baseline to Week 24 in Fasting Plasma Glucose (FPG) mmol/L
Description: Adjusted* mean change from baseline in fasting plasma glucose (FPG) achieved with saxagliptin 5 mg + metformin versus placebo + metformin at week 24 (Last Observation Carried Out (LOCF), Full Analysis set). FPG is a continuous measure, the change from baseline for each subject is calculated as the week 24 values minus the baseline value. *Adjusted for baseline FPG.
Time Frame: Baseline , Week 24
Population: as for outcome 1
Measure: Mean (Standard Error); unit: mmol/L
Arm/Group | Saxagliptin 5 mg + Metformin | Placebo + Metformin
Number analyzed (Participants) | 278 | 281
mmol/L
  Baseline | 8.57 (0.117) | 8.87 (0.137)
  Week 24 | 7.61 (0.117) | 8.30 (0.127)
  Adjusted Change from Baseline | -1.14 (0.114) | -0.58 (0.111)
Statistical Analysis 1: Comparison: Saxagliptin 5 mg + Metformin vs Placebo + Metformin; Test type: Superiority or Other; p < 0.0002, ANCOVA; Mean Difference (Net) = -0.56, 95% CI 2-sided [-0.85 to -0.26], Standard Error of Mean 0.149

3. Secondary Outcome: Absolute Change From Baseline to Week 24 in Fasting Plasma Glucose (FPG) mg/dL
Description: Adjusted* mean change from baseline in fasting plasma glucose (FPG) achieved with saxagliptin 5 mg + metformin versus placebo + metformin at week 24 (LOCF, Full Analysis set). FPG is a continuous measure, the change from baseline for each subject is calculated as the week 24 values minus the baseline value. *Adjusted for baseline FPG.
Time Frame: Baseline , Week 24
Population: as for outcome 1
Measure: Mean (Standard Error); unit: mg/dL
Arm/Group | Saxagliptin 5 mg + Metformin | Placebo + Metformin
Number analyzed (Participants) | 278 | 281
mg/dL
  Baseline | 154.54 (2.103) | 159.73 (2.467)
  Week 24 | 137.15 (2.116) | 149.54 (2.286)
  Adjusted Change from Baseline | -20.52 (2.051) | -10.42 (2.004)
Statistical Analysis 1: Comparison: Saxagliptin 5 mg + Metformin vs Placebo + Metformin; Test type: Superiority or Other; p < 0.0002, ANCOVA; Mean Difference (Net) = -10.10, 95% CI 2-sided [-15.37 to -4.83], Standard Error of Mean 2.684

4. Secondary Outcome: Change From Baseline in the Area Under the Curve (AUC) From 0 to 180 Minutes for Postprandial Glucose (PPG) During a Mixed Meal Tolerance Test (MMTT) in a Subgroup
Description: Adjusted* mean change from baseline in PPG AUC achieved with saxagliptin 5 mg + metformin versus placebo + metformin at week 24 (LOCF, Full Analysis set). Trapezoidal method was used to compute AUC under the 3 hour PPG curve. The change from baseline for each subject is calculated as the week 24 value minus the baseline value. *Adjusted for baseline PPG AUC.
Time Frame: Baseline , Week 24
Population: MMTT was measured on a subset of patients in China cohort only at baseline and Wk 24. Randomized participants who took at least 1 dose of double-blind treatment to be included in analysis: change from baseline to Wk 24 (LOCF), must have had a baseline and a post baseline data.
Measure: Mean (Standard Error); unit: mmol*min/L
Arm/Group | Saxagliptin 5 mg + Metformin | Placebo + Metformin
Number analyzed (Participants) | 113 | 111
mmol*min/L
  Baseline | 2355 (45.6) | 2427 (51.5)
  Week 24 | 2058 (44.4) | 2249 (46.9)
  Adjusted Change from Baseline | -315 (38.6) | -160 (39.0)
Statistical Analysis 1: Comparison: Saxagliptin 5 mg + Metformin vs Placebo + Metformin; Test type: Superiority or Other; p = 0.0052, ANCOVA; Mean Difference (Net) = -155, 95% CI 2-sided [-264 to -47], Standard Error of Mean 55.0

5. Secondary Outcome: Change From Baseline in the Area Under the Curve (AUC) From 0 to 180 Minutes for Postprandial Glucose (PPG) During a Mixed Meal Tolerance Test (MMTT) in a Subgroup
Description: Adjusted* mean change from baseline in PPG AUC achieved with saxagliptin 5 mg + metformin versus placebo+metformin at week 24 (LOCF, Full Analysis set). Trapezoidal method was used to compute AUC under the 3 hour PPG curve. The change from baseline for each subject is calculated as the week 24 value minus the baseline value. *Adjusted for baseline PPG AUC.
Time Frame: Baseline , Week 24
Population: as for outcome 4
Measure: Mean (Standard Error); unit: mg*min/dL
Arm/Group | Saxagliptin 5 mg + Metformin | Placebo + Metformin
Number analyzed (Participants) | 113 | 111
mg*min/dL
  Baseline | 42423 (821.9) | 43719 (927.3)
  Week 24 | 37071 (799.4) | 40521 (845.7)
  Adjusted Change from Baseline | -5673 (695.9) | -2871 (702.1)
Statistical Analysis 1: Comparison: Saxagliptin 5 mg + Metformin vs Placebo + Metformin; Test type: Superiority or Other; p = 0.0052, ANCOVA; Mean Difference (Net) = -2802, 95% CI 2-sided [-4753 to -852], Standard Error of Mean 989.8

6. Secondary Outcome: Proportion of Patients Achieving a Therapeutic Glycemic Response
Description: Proportion of participants achieving a therapeutic glycemic response, defined as having HbA1c < 7.0% for saxagliptin + metformin versus placebo + metformin at week 24
Time Frame: Baseline , Week 24
Population: Randomized participants who took at least 1 dose of double-blind treatment. To be included in analysis: change from baseline to Wk 24(LOCF) for efficacy, subjects must have had a baseline and at least 1 post baseline efficacy measurement.
Measure: Number; unit: Percentage of participants
Arm/Group | Saxagliptin 5 mg + Metformin | Placebo + Metformin
Number analyzed (Participants) | 275 | 279
Percentage of participants | 46.5 | 30.5
Statistical Analysis 1: Comparison: Saxagliptin 5 mg + Metformin vs Placebo + Metformin; Test type: Superiority or Other; p < 0.0001, ANCOVA; Mean Difference (Net) = 16.1, 95% CI 2-sided [8.0 to 24.0]

ADVERSE EVENTS:
Arm/Group | Saxagliptin 5 mg + Metformin | Placebo + Metformin
Serious Adverse Events (participants affected / at risk) | 8/283 | 3/287
Other Adverse Events (participants affected / at risk) | 19/283 | 13/287
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Saxagliptin 5 mg + Metformin (N=283) | Placebo + Metformin (N=287)
Anal Abscess (Infections and infestations) | 1 | 0
Appendicitis (Infections and infestations) | 1 | 0
Hepatitis B (Infections and infestations) | 1 | 0
Pulmonary Tuberculosis (Infections and infestations) | 1 | 0
Urinary Tract Infection (Infections and infestations) | 0 | 1
Ankle Fracture (Injury, poisoning and procedural complications) | 1 | 0
Clavicle Fracture (Injury, poisoning and procedural complications) | 1 | 0
Rib Fracture (Injury, poisoning and procedural complications) | 1 | 0
Cholecystitis Acute (Hepatobiliary disorders) | 1 | 0
Cerebral Infarction (Nervous system disorders) | 1 | 1
Diabetic Foot (Metabolism and nutrition disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Saxagliptin 5 mg + Metformin (N=283) | Placebo + Metformin (N=287)
Upper Respiratory Tract Infection (Infections and infestations) | 19 | 13

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Principal Investigator will provide AstraZeneca as soon as possible with preliminary data and drafts of proposed publications and disclosures, whether oral or in writing, with the proposed final manuscript. AZ shall have a period of 30 days from receipt of the proposed final manuscript for any publication or other disclosure to review it and may within such time require that submission for publication or disclosure of the manuscript be delayed.